CLINICAL TRIAL: NCT03133299
Title: A Study Evaluating Vitamin D in Allergic Bronchopulmonary Aspergillosis Complicating Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Consultant, Department of Pulmonary Medicine, Principal Investigator, Clinical Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pulm.Med/2017/002
Record Dates: First submitted 2017-04-21; First posted 2017-04-28 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Allergic Bronchopulmonary Aspergilloses
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Glucocorticoids; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid group (Active Comparator): Oral prednisolone 0.5 mg/kg/day for four weeks, 0.25 mg/kg/day for four weeks followed by 0.125 mg/kg/day for four weeks. Prednisolone will then be tapered by 5 mg every two weeks and discontinued. The total duration of glucocorticoids will be four months
  Interventions: Drug: Glucocorticoids
- Vitamin D plus Glucocorticoid group (Experimental): Oral vitamin D3 tablet, 60,000 IU weekly for 2 months (8 doses) along with Oral prednisolone 0.5 mg/kg/day for four weeks, 0.25 mg/kg/day for four weeks followed by 0.125 mg/kg/day for four weeks. Prednisolone will then be tapered by 5 mg every two weeks and discontinued. The total duration of glucocorticoids will be four months
  Interventions: Drug: Glucocorticoids; Drug: Vitamin D

INTERVENTIONS:
Drug: Glucocorticoids — Oral prednisolone for four months
Drug: Vitamin D — Oral vitamin D for two months
  Arms: Vitamin D plus Glucocorticoid group

SUMMARY:
Allergic bronchopulmonary aspergillosis (ABPA) is a immunological pulmonary disorder caused by hypersensitive reaction to spores of Aspergillus fumigatus. The prevalence of disease is about 1-2% in asthmatics and 2-15% in patients with cystic fibrosis. The interest in ABPA stems from the fact that the disease is glucocorticoid-sensitive and early treatment can prevent progression to end-stage lung disease. Recently anti-Th2 therapies have been suggested as treatment for ABPA. Vitamin D has been shown to suppress the Th2 responses and decrease the levels of Th2 interleukins. Hence, the investigators propose to assess the role of vitamin D in treating ABPA.

DETAILED DESCRIPTION:
Allergic bronchopulmonary aspergillosis (ABPA) is a immunological pulmonary disorder caused by hypersensitive reaction to spores of Aspergillus fumigatus. The prevalence of disease is about 1-2% in asthmatics and 2-15% in patients with cystic fibrosis. The interest in ABPA stems from the fact that the disease is glucocorticoid-sensitive and early treatment can prevent progression to end-stage lung disease.

Systemic steroids remain the mainstay of treatment in ABPA. Antifungal agents are also useful as they reduce fungal load. Newer therapies like omalizumab (anti immunoglobulin E [IgE] antibody), inhalational amphotericin and Anti Th2 therapies are being studied.

In pathogenesis of ABPA, there is heightened Th2 activity as a result of type 1 hypersensitive reaction to Aspergillus fumigatus and levels of Th2 cytokines like IL-3, IL-5 and IL-13 and IgE levels are increased in patients with ABPA compared with asthma patients without ABPA.

Recently anti Th2 therapies have been suggested as treatment for ABPA. Vitamin D has been shown to suppress the Th2 immunity and decrease the levels of Th2 interleukins. Hence, the investigators propose to assess the role of vitamin D in treatment of ABPA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ABPA as per the International Society for Human and Animal Mycology Working group criteria
* Treatment naïve

Exclusion Criteria:

* Failure to provide informed consent
* Enrollment in another trial of ABPA
* Pregnancy
* Creatinine more than or equal to 1.5 mg/dL
* Immunosuppressive states like chronic liver disease, chronic renal failure, cytotoxic therapy, uncontrolled diabetes mellitus and others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Decline in total IgE | Two months
  Total IgE at baseline and two months

SECONDARY OUTCOMES:
Decline in total IgE | Four months
  Total IgE at baseline and four months
Decline in total IgE | Six months
  Total IgE at baseline and six months
Th1/Th2 cytokines | Two months
  Th1 (IL-2 and interferon-gamma) and Th2 (IL4, IL5, IL10) cytokines at baseline and two months
Th1/Th2 cytokines | Four months
  Th1 (IL-2 and interferon-gamma) and Th2 (IL4, IL5, IL10) cytokines at baseline and four months
Th1/Th2 cytokines | Six months
  Th1 (IL-2 and interferon-gamma) and Th2 (IL4, IL5, IL10) cytokines at baseline and six months
Time to first exacerbation | One year
  The time to first exacerbation will be noted in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dodamani MH, Muthu V, Thakur R, Pal A, Sehgal IS, Dhooria S, Aggarwal AN, Garg M, Chakrabarti A, Agarwal R. A randomised trial of vitamin D in acute-stage allergic bronchopulmonary aspergillosis complicating asthma. Mycoses. 2019 Apr;62(4):320-327. doi: 10.1111/myc.12879. Epub 2019 Feb 5. PMID 30561849